CLINICAL TRIAL: NCT03799419
Title: Cognitive Bias Modification as an Adjunctive Treatment for Treatment-Refractory OCD
Brief Title: Cognitive Bias Modification for OCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Martha J Falkenstein, Staff Psychologist, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2017P002864
Record Dates: First submitted 2019-01-02; First posted 2019-01-10 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Obsessive-Compulsive Disorder; Obsessive-compulsive Disorders and Symptoms
Keywords: cognitive bias modification; interpretation bias; approach avoidance
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cognitive bias modification with treatment as usual (Experimental): Participants in this group will receive usual treatment in the program and 8 sessions of a computerized cognitive training targeting interpretation bias
  Interventions: Behavioral: Cognitive bias modification for interpretation bias
- Psychoeducation with treatment as usual (Sham Comparator): Participants in this group will receive usual treatment in the program and 8 sessions of psychoeducation
  Interventions: Behavioral: Psychoeducation
- Approach avoidance training with treatment as usual (Experimental): Participants in this group will receive usual treatment in the program and 8 sessions of a computerized cognitive training targeting automatic approach tendencies
  Interventions: Behavioral: Approach avoidance training
- Inactive sham approach avoidance training (Sham Comparator): Participants in this group will receive usual treatment in the program and 8 sessions of a sham approach avoidance training
  Interventions: Behavioral: Inactive sham approach avoidance training

INTERVENTIONS:
Behavioral: Cognitive bias modification for interpretation bias — Eight sessions of scenario-based CBM-I training for OCD will be administered, based on the widely-used paradigm of ambiguous scenario training developed by Mathews and Mackintosh (2000), in which participants are presented with scenarios that are ambiguous in whether or not they are threatening. Participants will complete a computer task consisting of a series of written scenarios designed to improve interpretation and attributional biases; these scenarios conclude with word fragments, which participants must fill in to resolve the ambiguity.
  Arms: Cognitive bias modification with treatment as usual
Behavioral: Psychoeducation — Eight sessions of psychoeducation will be administered, which will describe symptoms of anxiety, the nature of biased thinking in anxiety, and summarize common psychosocial as well as pharmacological treatments for anxiety. The sessions will provide relevant information but will not provide training in changing thinking styles.
  Arms: Psychoeducation with treatment as usual
Behavioral: Approach avoidance training — Eight sessions of this computerized training program will be used to train approach tendencies, following previously validated procedures (Najmi, Kuckertz, & Amir, 2010). During the training program, participants will view a series of these images and be prompted to push or pull a joystick according to prompts on the screen, instead of the content of the picture. Avoidance will be stimulated through both pushing away (images on the screen will decrease in size upon the joystick being pushed), and approach will be stimulated through pulling towards pictures (images will increase in size to simulate approach).
  Arms: Approach avoidance training with treatment as usual
Behavioral: Inactive sham approach avoidance training — Eight sessions of the approach avoidance training will be administered, however the percentage of push vs pull trials will be altered in this sham version of the training.
  Arms: Inactive sham approach avoidance training

SUMMARY:
This study will conduct the development and preliminary evaluation of Cognitive Bias Modification for Interpretation (CBM-I) and Approach Avoidance Training (AAT) as augmentations to treatment as usual for OCD and related disorders. CBM-I refers to computerized interventions designed to directly manipulate interpretation bias through repeated practice on a training task, thereby inducing cognitive changes in a relatively automatic or implicit manner. In AAT, automatic approach tendencies toward feared stimuli are re-trained. Specifically, this study will examine the feasibility, acceptability, and clinical outcomes associated with CBM-I and AAT.

Adults with obsessive compulsive disorder (OCD) and related disorders will be recruited from a treatment program for these disorders and participants will be randomly assigned to either receive: 1) eight sessions of CBM-I or eight sessions of psychoeducation as a control condition, or 2) AAT or eight sessions of an inactive (sham) version of the AAT training.

ELIGIBILITY:
Inclusion Criteria:

* Currently receiving treatment at the McLean Hospital OCD Institute
* For CBM-I condition only: report a score of at least 131 on the Obsessive Beliefs Questionnaire-44 upon admission to the OCD Institute
* For AAT condition only: endorse score of at least 7 on the DOCS subscale #1 (contamination subscale) upon admission to the OCD Institute
* Able to complete a computer task for 20 minutes
* Consent to main OCD Institute study protocol

Exclusion Criteria:

* Currently undergoing electroconvulsive therapy (ECT)
* Current symptoms of acute mania or psychosis
* A reported diagnosis at admission of a psychotic disorder
* History of traumatic brain injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2024-07-23 (Actual); Study Completion 2024-07-23 (Actual)

PRIMARY OUTCOMES:
Change in Average Score on Obsessive Beliefs Questionnaire | Weeks 0, 2, 4, and 8
  Measure of interpretation biases, specifically: Inflated Responsibility/Overestimation of Threat, Perfectionism/Intolerance of Uncertainty, and Importance/Control of Thoughts. 44-item self-report measure, items scored 1-7 and summed; greater scores indicate greater severity.

SECONDARY OUTCOMES:
Change in Average Score on Yale-Brown Obsessive Compulsive Scale | Weeks 0, 4, and 8
  Interviewer-rated measure of OCD symptoms. It is 19 items, with only items 1-10 scored (from 0-4). Total scores range from 0-40, with higher scores reflecting greater severity.
Change in Columbia-Suicide Severity Rating Scale | Weeks 0, 4, and 8
  An interviewer-rated assessment of retrospective suicidality as well as recent suicidal ideation and behavior. Minimum total score 0, maximum total score 5, higher total scores indicate more suicidal ideation and/or behavior.
Change in Suicide Implicit Association Test | Weeks 0, 2, and 4
  Computerized task which assesses implicit thoughts about self-injury, death, and suicide.
Change in Average Score on Depressive Symptom Index Suicidality Subscale. There are 4 items scored from 0-3 with greater numbers indicating greater severity. | Weeks 0, 1, 2, 3, and 4
  Self-report measure of suicidality
Credibility/Expectancy Questionnaire | Week 0
  Measure of treatment expectancy and rationale credibility in our study. The items are rated on 9-point scales, with a total score range of 3 to 27. Greater scores indicate greater expectations and perceptions of treatment credibility.
Exit Interview | Week 4
  This interview will be conducted by a member of the study staff to obtain participant feedback on satisfaction and how the intervention might be improved.
Change in Behavioral Approach Test | Weeks 0, 2, and 4
  Behavioral Approach Test (BAT) will be administered as a measure of OCD-related avoidance, based on previously validated procedures (Cougle et al., 2007; Amir, Kuckertz, & Najmi, 2013). Participants rate peak anxiety 0-100 for each step of approaching feared stimuli.
  Three different types of BAT will be implemented in order to measure avoidance with multiple types of contaminants, each with six steps on a hierarchy to be completed sequentially, providing a rating of anxiety 0-100 for each step.
Change in Average Score on Behavioral Inhibition/Behavioral Activation Scales | Weeks 0, 2, 4, and 8
  24-item measure of behavioral approach and behavioral avoidance, rated 1-4 and summed.
Dimensional Obsessive-Compulsive Scale | Weeks 0, 2, 4, and 8
  (DOCS; Abramowitz et al., 2010) participants with contamination fears will be identified by their DOCS contamination subscale score; the DOCS is part of the admission measures in the OCD Institute's main study protocol. Additionally, we will examine these scores as an outcome measure for contamination-related obsessions and compulsions. It includes 20 items and is rated 0-4.

CONTACTS AND LOCATIONS:
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States